CLINICAL TRIAL: NCT03623867
Title: Prevention of Metacarpophalangeal Joints Structure Damage in Patients With Psoriatic Arthritis Using Secukinumab
Brief Title: PsA Secukinumab XCT Structural Progression Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PsA secukinumab XCT study 2018
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Subject will be randomised into secukinumab or placebo group in 1:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Secukinumab (Experimental): Subject will received secukinumab 150mg at week 0-4, and once monthly till week 48
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Subject will received placebo 150mg at week 0-4, and once monthly till week 48
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Subject will take secukinumab once weekly in week 0-4, and once monthly till week 48
  Other Names: Cosentyx
  Arms: Secukinumab
Drug: Placebo — Subject will take placebo once weekly in week 0-4, and once monthly till week 48
  Arms: Placebo

SUMMARY:
Psoriatic arthritis is related with chronic inflammation and progressive radiographic damages, and it in turn lead to disability and loss in function-ability. Recent advance in treatment pathway through anti IL-17 gives promising clinical improvement. Yet, its effect on radiographic progression remains uncertain. This study aimed to ascertain the effect of secukinumab on structural progression in PsA by evaluation through high resolution peripheral quantative computed tomography (HRpqCT).

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic inflammatory joint disease associated with psoriasis. PsA is associated with distinctive clinical features including changes in skin and nails, peripheral arthritis, axial disease, dactylitis and enthesitis. Synovial inflammation in peripheral joints is the most prevalent feature of the disease ranging in severity from mild joint inflammation to disabling peripheral arthritis [1]. Within 2 years of diagnosis, radiological erosions were developed in 47% of the patients [2]. Without proper monitoring and treatment, it will lead to significant structure damage and loss of physical function, and even arthritis mutilans, which is the most severe destructive form of PsA [3]. Prevention of structural damage is one of the primary goals of treating PsA patients to maximise health-related quality of life [4].

Detection of bone erosions in PsA patients is usually achieved by conventional radiographs although the sensitivity is low [5]. High-resolution peripheral quantitative CT (HR-pQCT) is a novel technique for detailed bone microstructure analysis with high reproducibility in assessing bony erosions [6]. With its high spatial resolution of 130 μm, HR-pQCT exhibited a higher sensitivity in detecting erosion compared with radiograph and magnetic resonance imaging (MRI) [7]. Recently, Finzel et al. described an indirect method to assess volume based on measurements of the width and depth of the erosions using HR-pQCT [8]. Quantitative measurement of erosion volume can also be achieved [6]. Using this method, erosion repair under biological disease-modifying antirheumatic drugs (DMARDs) treatment has been demonstrated in patients with rheumatoid arthritis (RA) [8, 9]. Bone apposition at the margin of erosions (osteosclerosis) with the formation of a new cortical lining was associated with a decrease in erosion depth or width, which may indicate either periosteal or endosteal repair processes [8, 9]. Valid measurement of erosion volume using HR-pQCT will facilitate the testing of treatments that may help to heal erosion. Decrease in erosion volume and the presence of osteosclerosis on HR-pQCT could be promising markers for erosion healing.

Interleukin 17 (IL-17) is a proinflammatory cytokine which produced by type 17 helper T cells (Th17). It is now considered to be a key cytokine in the pathogenesis of a number of autoimmune disorders in humans including PsA [10]. IL-17 was also reported to be associated with the presence of joint erosion [11]. Recently, secukinumab, an anti-interleukin-17A monoclonal antibody, was reported to be effective in reducing disease activity and decreased the rate of radiographic joint damage compared with placebo [12]. However, whether healing of erosion could occur in PsA has never been evaluated.

On the other hand, osteophytes formation at the entheseal regions of the joints in PsA is distinctive feature compared with RA [13]. The formation of osteophytes is tightly regulated by anabolic pathways, which resembles the pathogenesis of new bone formation in ankylosing spondylitis (AS). Tumor necrosis factor (TNF) inhibition was unable to halt the structural progression in AS patients [14-16], it also lacked efficacy in stopping the progression of osteophytes in PsA patients [17]. Inhibition of IL-17 by secukinumab was effective in the treatment of both AS [18] and PsA [12]. Secukinumab also decreased the rate of radiographic joint damage regarding to erosion and joint space narrowing [12]. However, it is unknown if it has any effect in the progression of osteophytes. In an animal model, although over-expression of IL-17 alone failed to induce entheseal and periosteal bone formation, inhibition of IL-17 leaded to significant reduction of such bone formation in an IL-23 overexpression model [19]. Moreover, IL-17A accelerates bone formation by stimulating the proliferation and osteoblastic differentiation of mesenchymal progenitor cells after injury [20]. It is worth exploring if secukinumab could prevent the progression of osteophytes in PsA patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. without severe deformity in MCP joints which would influence the longitudinal assessment of HR-pQCT;
3. with active disease, which is defined as three or more than tender joints and three or more than swollen joints, despite previous treatment with nonsteroidal anti-inflammatory drugs, disease-modifying antirheumatic drugs.

Exclusion Criteria:

1. limited in ability to perform usual self-care, vocational, and avocational activities;
2. pregnancy;
3. previous therapy with biologic;
4. the presence of active inflammatory diseases other than PsA;
5. active infection in 2 weeks before randomization or a history of ongoing, chronic, or recurrent infections including tuberculosis;
6. history of hepatitis B & C;
7. history of malignant disease within the past 5 years (excluding basal cell carcinoma or actinic keratosis, in-situ cervical cancer, or non-invasive malignant colon polyps);
8. contraindications to secukinumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Difference in changes in the volume of erosions on metacarpophalangeal joints (MCP) 2-4 measured by HR-pQCT at 24 weeks between secukinumab and placebo group | 24 weeks
  The erosion volume will be calculated from HR-pQCT images
Difference in changes in the volume of erosions on metacarpophalangeal joints (MCP) 2-4 measured by HR-pQCT at 48 weeks between secukinumab and placebo group | 48 weeks
  The erosion volume will be calculated from HR-pQCT images

SECONDARY OUTCOMES:
The percentage of erosions with healing determined using HR-pQCT on MCP 2-4 | 24 weeks
  Erosion healing is defined as a decrease in erosion volume of ≥0.4 mm3 from baseline, and the presence of grade 2 osteosclerosis at the margin of erosion
The percentage of erosions with healing determined using HR-pQCT on MCP 2-4 | 48 weeks
  Erosion healing is defined as a decrease in erosion volume of ≥0.4 mm3 from baseline, and the presence of grade 2 osteosclerosis at the margin of erosion
Changes in depth and width of erosion using HR-pQCT | 24 weeks
  The erosion volume will be calculated from HR-pQCT images
Changes in depth and width of erosion using HR-pQCT | 48 weeks
  The erosion volume will be calculated from HR-pQCT images
Marginal osteosclerosis using HR-pQCT | 24 weeks
  The marginal osteosclerosis will be calculated from HR-pQCT images
Marginal osteosclerosis using HR-pQCT | 48 weeks
  The marginal osteosclerosis will be calculated from HR-pQCT images
Changes in the height of osteophytes using HR-pQCT | 24 weeks
  The height of osteophytes will be analysed from HR-pQCT images
Changes in the height of osteophytes using HR-pQCT | 48 weeks
  The height of osteophytes will be analysed from HR-pQCT images
Changes in joint space volume using HR-pQCT | Week 24
  HR-pQCT measures the joint space volume
Changes in joint space volume using HR-pQCT | Week 48
  HR-pQCT measures the joint space volume

OTHER OUTCOMES:
Changes in HAQ (Health Assessment Questionnaire) | Week 24
  HAQ (0-3) assessing functional disability, with higher score representing higher functional disability.
Changes in HAQ (Health Assessment Questionnaire) | Week 48
  HAQ (0-3) assessing functional disability, with higher score representing higher functional disability.
Changes in patient reported outcome (SF-36) | Week 48
  SF-36 is a questionnaire representing subject's physical & mental well being ranging from 0-100, with 100 representing better outcome.
Changes in patient reported outcome (SF-36) | Week 24
  SF-36 is a questionnaire representing subject's physical & mental well being ranging from 0-100, with 100 representing better outcome.
Changes in Psoriatic Arthritis Impact of Disease (PsAID) | Week 24
  PsAID (0-12) measures the impact of PsA in patients with lower score representing better QoL
Changes in Psoriatic Arthritis Impact of Disease (PsAID) | Week 48
  PsAID (0-12) measures the impact of PsA in patients with lower score representing better QoL
Changes in van der Heijde-Sharp score on radiograph at 48 weeks | 48 weeks
  The van der Heijde-sharp score assess erosion (0-528) and joint space narrowing (0-208) in x-ray, which higher score represent higher radiographic damages

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mortezavi M, Thiele R, Ritchlin C. The joint in psoriatic arthritis. Clin Exp Rheumatol. 2015 Sep-Oct;33(5 Suppl 93):S20-5. Epub 2015 Oct 15. PMID 26472472
- [Background] Kane D, Stafford L, Bresnihan B, FitzGerald O. A prospective, clinical and radiological study of early psoriatic arthritis: an early synovitis clinic experience. Rheumatology (Oxford). 2003 Dec;42(12):1460-8. doi: 10.1093/rheumatology/keg384. Epub 2003 Oct 1. PMID 14523223
- [Background] Acosta Felquer ML, FitzGerald O. Peripheral joint involvement in psoriatic arthritis patients. Clin Exp Rheumatol. 2015 Sep-Oct;33(5 Suppl 93):S26-30. Epub 2015 Oct 15. PMID 26471860
- [Background] Gossec L, Smolen JS, Ramiro S, de Wit M, Cutolo M, Dougados M, Emery P, Landewe R, Oliver S, Aletaha D, Betteridge N, Braun J, Burmester G, Canete JD, Damjanov N, FitzGerald O, Haglund E, Helliwell P, Kvien TK, Lories R, Luger T, Maccarone M, Marzo-Ortega H, McGonagle D, McInnes IB, Olivieri I, Pavelka K, Schett G, Sieper J, van den Bosch F, Veale DJ, Wollenhaupt J, Zink A, van der Heijde D. European League Against Rheumatism (EULAR) recommendations for the management of psoriatic arthritis with pharmacological therapies: 2015 update. Ann Rheum Dis. 2016 Mar;75(3):499-510. doi: 10.1136/annrheumdis-2015-208337. Epub 2015 Dec 7. PMID 26644232
- [Background] Poggenborg RP, Bird P, Boonen A, Wiell C, Pedersen SJ, Sorensen IJ, Madsen OR, Slot O, Moller JM, Boyesen P, Hasselquist M, Ostergaard M. Pattern of bone erosion and bone proliferation in psoriatic arthritis hands: a high-resolution computed tomography and radiography follow-up study during adalimumab therapy. Scand J Rheumatol. 2014;43(3):202-8. doi: 10.3109/03009742.2013.835865. Epub 2013 Dec 19. PMID 24354412
- [Background] Fouque-Aubert A, Boutroy S, Marotte H, Vilayphiou N, Bacchetta J, Miossec P, Delmas PD, Chapurlat RD. Assessment of hand bone loss in rheumatoid arthritis by high-resolution peripheral quantitative CT. Ann Rheum Dis. 2010 Sep;69(9):1671-6. doi: 10.1136/ard.2009.114512. Epub 2010 Jun 4. PMID 20525847
- [Background] Srikhum W, Virayavanich W, Burghardt AJ, Yu A, Link TM, Imboden JB, Li X. Quantitative and semiquantitative bone erosion assessment on high-resolution peripheral quantitative computed tomography in rheumatoid arthritis. J Rheumatol. 2013 Apr;40(4):408-16. doi: 10.3899/jrheum.120780. Epub 2013 Feb 15. PMID 23418386
- [Background] Finzel S, Rech J, Schmidt S, Engelke K, Englbrecht M, Schett G. Interleukin-6 receptor blockade induces limited repair of bone erosions in rheumatoid arthritis: a micro CT study. Ann Rheum Dis. 2013 Mar;72(3):396-400. doi: 10.1136/annrheumdis-2011-201075. Epub 2012 May 14. PMID 22586162
- [Background] Finzel S, Rech J, Schmidt S, Engelke K, Englbrecht M, Stach C, Schett G. Repair of bone erosions in rheumatoid arthritis treated with tumour necrosis factor inhibitors is based on bone apposition at the base of the erosion. Ann Rheum Dis. 2011 Sep;70(9):1587-93. doi: 10.1136/ard.2010.148395. Epub 2011 May 27. PMID 21622765
- [Background] Miossec P, Korn T, Kuchroo VK. Interleukin-17 and type 17 helper T cells. N Engl J Med. 2009 Aug 27;361(9):888-98. doi: 10.1056/NEJMra0707449. No abstract available. PMID 19710487
- [Background] Menon B, Gullick NJ, Walter GJ, Rajasekhar M, Garrood T, Evans HG, Taams LS, Kirkham BW. Interleukin-17+CD8+ T cells are enriched in the joints of patients with psoriatic arthritis and correlate with disease activity and joint damage progression. Arthritis Rheumatol. 2014 May;66(5):1272-81. doi: 10.1002/art.38376. PMID 24470327
- [Background] Mease PJ, McInnes IB, Kirkham B, Kavanaugh A, Rahman P, van der Heijde D, Landewe R, Nash P, Pricop L, Yuan J, Richards HB, Mpofu S; FUTURE 1 Study Group. Secukinumab Inhibition of Interleukin-17A in Patients with Psoriatic Arthritis. N Engl J Med. 2015 Oct;373(14):1329-39. doi: 10.1056/NEJMoa1412679. PMID 26422723
- [Background] Finzel S, Englbrecht M, Engelke K, Stach C, Schett G. A comparative study of periarticular bone lesions in rheumatoid arthritis and psoriatic arthritis. Ann Rheum Dis. 2011 Jan;70(1):122-7. doi: 10.1136/ard.2010.132423. Epub 2010 Oct 11. PMID 20937672
- [Background] van der Heijde D, Salonen D, Weissman BN, Landewe R, Maksymowych WP, Kupper H, Ballal S, Gibson E, Wong R; Canadian (M03-606) study group; ATLAS study group. Assessment of radiographic progression in the spines of patients with ankylosing spondylitis treated with adalimumab for up to 2 years. Arthritis Res Ther. 2009;11(4):R127. doi: 10.1186/ar2794. Epub 2009 Aug 24. PMID 19703304
- [Background] van der Heijde D, Landewe R, Baraliakos X, Houben H, van Tubergen A, Williamson P, Xu W, Baker D, Goldstein N, Braun J; Ankylosing Spondylitis Study for the Evaluation of Recombinant Infliximab Therapy Study Group. Radiographic findings following two years of infliximab therapy in patients with ankylosing spondylitis. Arthritis Rheum. 2008 Oct;58(10):3063-70. doi: 10.1002/art.23901. PMID 18821688
- [Background] van der Heijde D, Landewe R, Einstein S, Ory P, Vosse D, Ni L, Lin SL, Tsuji W, Davis JC Jr. Radiographic progression of ankylosing spondylitis after up to two years of treatment with etanercept. Arthritis Rheum. 2008 May;58(5):1324-31. doi: 10.1002/art.23471. PMID 18438853
- [Background] Finzel S, Kraus S, Schmidt S, Hueber A, Rech J, Engelke K, Englbrecht M, Schett G. Bone anabolic changes progress in psoriatic arthritis patients despite treatment with methotrexate or tumour necrosis factor inhibitors. Ann Rheum Dis. 2013 Jul;72(7):1176-81. doi: 10.1136/annrheumdis-2012-201580. Epub 2012 Aug 21. PMID 22915620
- [Background] Baeten D, Sieper J, Braun J, Baraliakos X, Dougados M, Emery P, Deodhar A, Porter B, Martin R, Andersson M, Mpofu S, Richards HB; MEASURE 1 Study Group; MEASURE 2 Study Group. Secukinumab, an Interleukin-17A Inhibitor, in Ankylosing Spondylitis. N Engl J Med. 2015 Dec 24;373(26):2534-48. doi: 10.1056/NEJMoa1505066. PMID 26699169
- [Background] Sherlock JP, Joyce-Shaikh B, Turner SP, Chao CC, Sathe M, Grein J, Gorman DM, Bowman EP, McClanahan TK, Yearley JH, Eberl G, Buckley CD, Kastelein RA, Pierce RH, Laface DM, Cua DJ. IL-23 induces spondyloarthropathy by acting on ROR-gammat+ CD3+CD4-CD8- entheseal resident T cells. Nat Med. 2012 Jul 1;18(7):1069-76. doi: 10.1038/nm.2817. PMID 22772566
- [Background] Ono T, Okamoto K, Nakashima T, Nitta T, Hori S, Iwakura Y, Takayanagi H. IL-17-producing gammadelta T cells enhance bone regeneration. Nat Commun. 2016 Mar 11;7:10928. doi: 10.1038/ncomms10928. PMID 26965320

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03623867/Prot_SAP_001.pdf